CLINICAL TRIAL: NCT00356317
Title: A Culturally Based Family Therapy for Schizophrenia
Brief Title: Culturally Based Family Therapy for Improving Treatment Outcome for People With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amy Weisman, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH071250 (NIH); R34MH071250 (NIH); DSIR 83-ATAP
Record Dates: First submitted 2006-07-21; First posted 2006-07-25 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Schizophrenia
Keywords: Culture; Family; Therapy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive a 15-week family therapy
  Interventions: Behavioral: Culturally informed therapy for schizophrenia (CIT-S)
- 2 (Active Comparator): Participants will receive a 3-week family therapy (treatment as usual)
  Interventions: Behavioral: Psychoeducation treatment as usual

INTERVENTIONS:
Behavioral: Culturally informed therapy for schizophrenia (CIT-S) — This family therapy consists of 15 video-taped, therapy sessions, each lasting approximately 75 minutes. The 15-session treatment will be broken down into five segments (each lasting approximately three sessions) with the following goals: 1) Fortify a strong sense of family unity; 2) educate about schizophrenia; 3) foster adaptive use of cultural, spiritual and/or existential beliefs in conceptualizing and coming to terms with schizophrenia; 4) teach effective communication training techniques; and 5) and teach useful problem solving strategies.
  Arms: 1
Behavioral: Psychoeducation treatment as usual — This family therapy consists of three weekly sessions focusing on education about schizophrenia.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of a culturally based family therapy intervention in improving treatment outcome in people with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a disabling mental disorder that affects approximately 1% of the population worldwide. People with schizophrenia frequently experience hallucinations, delusions, disordered thinking, movement disorders, emotional numbness, social withdrawal, and cognitive deficits. These symptoms can hinder a person's ability to perform everyday functions, such as hold a job and maintain normal social relationships. When combined with medication, family-oriented therapy interventions have been beneficial for people with schizophrenia. There are few programs, however, that are tailored to the needs of minorities. With the rising number of minority populations in the U.S., it is important to develop psychotherapy interventions that are designed specifically for these groups. This study will evaluate the effectiveness of a culturally based family therapy intervention in improving treatment outcome in people with schizophrenia.

Participants in this 12-month, open label study will first attend a 2-hour screening visit, at which information will be gathered regarding coping styles, spirituality, and expressed emotion. Participants will then be randomly assigned to receive either culturally based therapy or treatment as usual. Although the culturally based therapy will be tailored to the needs and values of Hispanics, people who are not Hispanic will not be excluded. The culturally based therapy will entail 15 weekly therapy sessions, which will focus on family unity, psychoeducation, spirituality, communication skills, and problem-solving. The group receiving treatment as usual will attend 3 weekly psychoeducation sessions that will focus on informing participants about schizophrenia. Outcomes for both groups will be assessed upon completion of treatment and at follow-up visits at Months 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

For participants with schizophrenia or schizoaffective disorder:

* Diagnosis of schizophrenia or schizoaffective disorder
* Currently taking medication
* 18 or older

For all participants:

* Two or more family members, including patient, are available for participation (therapy can be conducted if patient is not available, as long as two other family members are interested in participating)
* Family members must be at least 13 years old

Exclusion Criteria:

* N/A

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Schizophrenia symptom severity | Measured immediately post-treatment and at Months 6 and 12

SECONDARY OUTCOMES:
Symptoms of depression, anxiety, and stress | Measured immediately post-treatment and at Months 6 and 12
Family functioning | Measured immediately post-treatment and at Months 6 and 12
Cultural Identity | Measured immediately post-treatment and at Months 6 and 12
Coping styles | Measured immediately post-treatment and at Months 6 and 12
Religiosity/Spirituality | Measured immediately post-treatment and at Months 6 and 12
Alcohol and Drug Use | Measured immediately post-treatment and at Months 6 and 12
Knowledge and knowledge about schizophrenia | Measured immediately post-treatment and at Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Amy Weisman, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

REFERENCES:
- [Background] Weisman A, Duarte E, Koneru V, Wasserman S. The development of a culturally informed, family-focused treatment for schizophrenia. Fam Process. 2006 Jun;45(2):171-86. doi: 10.1111/j.1545-5300.2006.00089.x. PMID 16768017